CLINICAL TRIAL: NCT04207944
Title: Preventing an Incurable Disease: The Prevention of Progression to Pancreatic Cancer Trial (The 3P-C Trial)
Brief Title: The Prevention of Progression to Pancreatic Cancer Trial (The 3P-C Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Johns Hopkins University (Other); Massachusetts General Hospital (Other); Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00103684; 1R01CA235677-01A1 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: IPMN; IPMN, Pancreatic
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms | interventions — Sulindac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sulindac (Experimental): Patients will be randomized to receive standard radiographic/endoscopic surveillance plus sulindac. The sulindac starting dose is 200 mg by mouth 2x daily. Patients will continue drug for 3 years during follow-up.
  Interventions: Drug: Sulindac 400 MG
- Placebo (Placebo Comparator): Patients will be randomized to receive standard radiographic/endoscopic surveillance plus placebo. Patients will continue placebo for 3 years during follow-up.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sulindac 400 MG — Patients will be randomized to receive standard radiographic/endoscopic surveillance plus sulindac. The sulindac starting dose is 200 mg by mouth 2x daily. Randomization will be performed at Duke and stratified by (1) the presence of high-grade dysplasia on the operative pathologic report and (2) the use of metformin at the time of enrollment. Patients will be provided the study drugs by a Duke, MSK, MGH, or JHH pharmacist. Patients will continue drug/placebo for 3 years during follow-up.
  Arms: Sulindac
Other: Placebo — Patients will be randomized to receive standard radiographic/endoscopic surveillance plus sulindac. The sulindac starting dose is 200 mg by mouth 2x daily. Randomization will be performed at Duke and stratified by (1) the presence of high-grade dysplasia on the operative pathologic report and (2) the use of metformin at the time of enrollment. Patients will be provided the study drugs by a Duke, MSK, MGH, or JHH pharmacist. Patients will continue drug/placebo for 3 years during follow-up.
  Arms: Placebo

SUMMARY:
This is a multi-center randomized double-blind placebo controlled trial of patients with high-risk intraductal papillary mucinous neoplasms (IPMNs) of the pancreas. The primary objective is to evaluate the effect of sulindac on the presence or absence of progression of IPMN after up to 3 years of treatment.

Patients without contraindications will be considered to be eligible and will be required to have a cross-sectional imaging study of the pancreas by CT scan or MRI within 3 months of study entry to document residual IPMNs and to rule out any evidence of pancreatic cancer. Patients will be randomized to receive either sulindac (200 mg p.o. BID) plus standard radiographic and endoscopic surveillance or placebo plus standard radiographic and endoscopic surveillance. Randomization will be stratified by (1) whether the patient had high-grade dysplasia identified in the initial resection specimen (resected patients only) and (2) whether the patient is taking metformin at the time of randomization.

DETAILED DESCRIPTION:
This is a phase 2 multicenter, randomized, double-blind, placebo-controlled clinical trial of patients who have high-risk intraductal papillary mucinous neoplasms (IPMN) of the pancreas. Patients will be randomized in a 1:1 fashion and stratified by whether the patient had high-grade dysplasia (yes vs. no vs. no resection) identified in the initial resection specimen (for resected subjects), and whether or not the patient is taking metformin at the time of randomization. Patients will be required to have undergone an MRI or CT angiogram for IPMN active surveillance in accordance with the standard practice at the enrolling institution within 3 months of study entry. The CT imaging study will be used to document baseline IPMN characteristics and to ensure that there is no evidence of a preexisting pancreatic cancer.

Following randomization, patients will take the study drug or placebo twice daily for up to 3 years. Both the study drug arm and the placebo arm will undergo standard laboratory, radiographic, and endoscopic assessment for IPMN progression. Every 6 months, patients will undergo assessment of serum CMP, CBC, and CA19-9. EUS will be performed 6 months after randomization (+/- 4 weeks) and then annually. CT or MRI will be performed 1 year after randomization (+/- 4 weeks) and then annually. The intent of these timings is to have the EUS and CT/MRI be on an alternating 6-month schedule per standard of care.

Patients, nurses, and physicians will be blinded to the randomization. Study drug will be provided to patients in the outpatient clinic or mailed to their home. Pill diaries will be provided at the time that the study drugs are given and will be evaluated every 6 months, at the time of routine follow-up.

Safety and efficacy will be assessed throughout the treatment period. Assessment for study drug complications will be made by phone call every other month (in between routine follow-up) and at routine follow-up every 6 months by the attending surgeon or designee, until the end of the study. If a complication is identified, the study drug will be discontinued. Patient evaluations will be scheduled bi-annually for the primary endpoint and off-schedule evaluations may be made to address symptoms or clinical concerns as they arise.

The investigators plan to accrue 100 patients and will follow all patients for up to 3 additional years until protocol defined progression or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or woman between the ages of 21 and 85 (inclusive) years.
2. Subject has high-risk IPMN as defined below.

   1. Patient (previously resected) has undergone partial pancreatectomy for non-invasive IPMN AND has new or residual cyst(s) > 1 cm and/or
   2. Patient (not previously resected) has a radiographic lesion of the pancreas consistent with IPMN as documented by: Cyst fluid CEA > 192 ng/ml OR presence of GNAS or RNF 43 mutation noted in cyst fluid OR MRI imaging confirmation of "likely", "probable" or "confirmed" communication with main pancreatic duct

   AND at least one of the following worrisome features:
   * Cyst > 2.5 cm
   * Thickened/enhancing cyst walls
   * Main pancreatic duct > 5mm
   * Abrupt change in caliber of pancreatic duct with distal atrophy
3. Subjects has ECOG of 0-2
4. Subject is medically fit to undergo EUS.
5. Female subjects who are of childbearing potential or are capable of becoming pregnant must be willing to use appropriate methods of contraception for the length of the study.
6. Subject is able to provide written informed consent.

Exclusion Criteria:

1. Subject has pathologic evidence of pancreatic adenocarcinoma.
2. Subject takes a systemic corticosteroid or NSAID more than 3 times per week.
3. Subject has a known history of or currently existing allergy to NSAIDs, aspirin induced asthma, gastric ulcers, non-iatrogenic intestinal perforation, or gastrointestinal bleeding from NSAID usage for which intervention was required..
4. Subject has an ongoing history of renal insufficiency (eGFR <50 mL/minute/1.73 m2), cardiovascular disease, gastrointestinal disorder, or any other condition that serves as a contraindication to the use of sulindac in the opinion of the treating investigator.
5. Myocardial infarction or coronary artery bypass grafting within six months of study entry.
6. Diagnosis of Congestive Heart Failure.
7. Severe adverse drug reaction to contrast agents that cannot be managed with routine premedication prior to imaging.
8. Diagnosis for (other) prior malignancy (except in situ and non-melanoma skin cancers) and are actively receiving antineoplastic or immuno therapy within 90 days of randomization.
9. History of medical procedure that would prevent an endoscopic ultrasound from being performed (such as Roux-en-Y, prior total gastrectomy).
10. Subject is lactating or pregnant.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percent of patients with IPMN progression as measured by a composite of several indicators | 3 years
  Patients will be determined to have progressed if they have:
  1. New cystic lesion(s) of the pancreas >1 cm in diameter (or initial lesion(s) <5 mm that are now >1cm),
  2. Doubling of the diameter of any preexisting cyst initially measuring ≥5 mm
  3. Increase in diameter of the main pancreatic duct by >3mm
  4. Pancreatic resection
  5. The development of pancreatic adenocarcinoma

SECONDARY OUTCOMES:
Percent of patients with cyst progression as measured by radiographic images | 3 years
  1. All initial and follow-up radiographic imaging will be quantitatively assessed for radiographic changes associated with progression. Utilizing a recently described radiomics approach to the evaluation of imaging in patients with IPMN, the investigators will further explore the set of 256 imaging features that broadly describe variation in radiographic enhancement patterns (i.e. heterogeneity). Using image analysis techniques, the investigators will derive quantitative measurements of the cyst wall and will determine the presence and degree of solid enhancing component suggestive of malignancy.

OTHER OUTCOMES:
Percent of patients with Inflammatory Marker Progression | 3 years
  2. Cyst fluid obtained at the time of annual EUS or surgical resection will be used to determine whether cyst fluid inflammatory marker analysis can identify progression. Antibody bead array analysis will be used to assess whether previously developed biomarker models for high-risk IPMN (IL-4/sFASL and MMP-9/CA72-4) can identify patients with an increased risk of radiographic progression. Archival tissue will be collected to validate cyst fluid analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Allen, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data will only be shared through publication.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT04207944/ICF_000.pdf